CLINICAL TRIAL: NCT00372567
Title: A Phase IIIB, Randomized, Active Controlled Open-Label Study Of Sunitinib (Sutent) 37.5 Mg Daily Vs Imatinib Mesylate 800 Mg Daily In The Treatment Of Patients With Gastrointestinal Stromal Tumors (GIST) Who Have Had Progressive Disease While On 400 Mg Daily Of Imatinib
Brief Title: Safety And Effectiveness Of Daily Dosing With Sunitinib Or Imatinib In Patients With Gastrointestinal Stromal Tumors
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181112
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2010-12-31 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Sunitinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: sunitinib malate
- B (Active Comparator)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: sunitinib malate — 37.5 mg daily
  Other Names: Sutent
  Arms: A
Drug: imatinib mesylate — 800mg daily
  Arms: B

SUMMARY:
A phase IIIb study of patients with gastrointestinal stromal tumors who have had progressive disease while on 400 mg imatinib. Patients will be randomly assigned to either sunitinib 37.5 mg daily or imatinib 800 mg daily. This study will find out the benefits and potential side effects of taking sunitinib or imatinib for approximately one year.

DETAILED DESCRIPTION:
The study prematurely discontinued on July 27, 2009 due to poor recruitment and operational futility as a result of changes in clinical practice. There were no safety or efficacy concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastrointestinal stromal tumors whose disease has progressed on imatinib 400 mg daily.

Exclusion Criteria:

* Current treatment with any chemotherapy other than imatinib.
* Current treatment with any dose of imatinib other than 400 mg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- United States (6):
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
- Germany (2):
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hamburg
- Hong Kong (3):
  - Pfizer Investigational Site, Lai Chi Kok, Kowloon
  - Pfizer Investigational Site, Tuenmen, New Territories
  - Pfizer Investigational Site, Hong Kong
- Italy (3):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, San Giovanni Rotondo
- Pfizer Investigational Site, Seoul, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Valencia, Valencia
- United Kingdom (4):
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181112&StudyName=Safety%20And%20Effectiveness%20Of%20Daily%20Dosing%20With%20Sunitinib%20Or%20Imatinib%20In%20Patients%20With%20Gastrointestinal%20Stromal%20Tumors%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants were enrolled in a lead-in Phase 1 safety sub-study, all of whom received Sunitinib 37.5 milligram (mg) 24 hours after the last dose of imatinib. No efficacy evaluations were planned/conducted for this sub-study.
Groups:
- Sunitinib (Phase 3): Starting dose of 37.5 mg once daily (QD) on Days 1, 7, and 14 for each cycle. Dose adjustments, if needed, included a reduction to 25 mg QD or an escalation to 50 mg QD.
- Imatinib: Starting dose of 800 mg QD on Days 1, 7, and 14 for each cycle. Dose adjustments, if needed, included a reduction to 600 mg QD.
- Sunitinib (Phase 1): Single 37.5 mg dose administered 24 hours after the last dose of imatinib
Period: Phase 1 Sub-study
Arm/Group | Sunitinib (Phase 3) | Imatinib | Sunitinib (Phase 1)
Started | 0 | 0 | 12
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 0
Period: Phase 3 Study
Arm/Group | Sunitinib (Phase 3) | Imatinib | Sunitinib (Phase 1)
Started | 31 | 26 | 12
Received Treatment | 31 | 25 | 12
Completed | 0 | 0 | 0
Not Completed | 31 | 26 | 12
Not completed — Adverse Event | 5 | 1 | 1
Not completed — Death | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Objective progression or relapse | 10 | 13 | 4
Not completed — Global deterioration of health status | 0 | 1 | 0
Not completed — Other | 2 | 2 | 1
Not completed — study terminated by sponsor | 13 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib (Phase 3) | Imatinib | Sunitinib (Phase 1) | Total
Number analyzed (Participants) | 31 | 26 | 12 | 69
Age, Customized [Number; unit: participants]
  less than 65 years | 19 | 17 | 7 | 43
  greater than or equal to 65 years | 12 | 9 | 5 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 5 | 27
  Male | 20 | 15 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time from randomization to the first documentation of tumor progression or death due to any cause in the absence of documented tumor progression, whichever was earlier.
Time Frame: Baseline, Week 5, and every 8 weeks until Year 2
Population: Intention to treat (ITT): all participants in Main Study (Phase 3) who were randomized, regardless of whether the participant received any drug or received a different drug from that to which they were randomized. Number of participants analyzed: participants who had a PFS event (progressive disease or death).
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Sunitinib: Starting dose of 37.5 mg once daily (QD) on Days 1, 7, and 14 for each cycle. Dose adjustments, if needed, included a reduction to 25 mg QD or an escalation to 50 mg QD.
Arm/Group | Sunitinib | Imatinib
Number analyzed (Participants) | 13 | 15
Months | 8.6 [5.7 to 9.0] | 6.4 [4.5 to 15.7]
Statistical Analysis 1: Comparison: Sunitinib vs Imatinib; No hypothesis tested; Test type: Superiority or Other; Cox Proportional Hazards Model; Model stratified by previous imatinib treatment status (less than 6 months of treatment with imatinib and greater than or equal to 6 months); Hazard Ratio (HR) = 1.040, 95% CI 2-sided [0.484 to 2.235]

2. Secondary Outcome: Overall Survival (OS)
Description: Time from date of randomization to the date of death. In the absence of confirmation of death, survival time was censored to the last date the participant was known to be alive.
Time Frame: Baseline up to 2 years
Population: ITT
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 31 | 26
Months | 12.9 [10.7 to 12.9] | NA [NA to NA] — The estimate of median OS in the Imatinib Treatment Arm was not available (NA) because data was not mature.
Statistical Analysis 1: Comparison: Sunitinib (Phase 3) vs Imatinib; Test type: Superiority or Other; Cox Proportional Hazards Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.818, 95% CI 2-sided [0.640 to 12.41]

3. Secondary Outcome: Time to Pain Relief Response (TTPR)
Description: Pain relief response defined as a 50 percent (%) or more reduction in the McGill Pain Questionaire - Present Pain Intensity (MPQ-PPI) score (0=no pain to 5=excruciating pain) and/or analgesic use from baseline for at least 3 consecutive weeks. Analgesic use scores were based on 1 point per non narcotic dose of medication and 4 points per dose of narcotic medication.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 31 | 26
Days | 34.0 [11.0 to 57.0] | 22.0 [8.0 to 113.0]

4. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF included death for any reason, treatment termination due to intolerable toxicity, or withdrawal of consent, whichever occurred first.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT; Number of participants analyzed: participants with treatment failure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 16 | 17
Months | 8.2 [5.5 to 9.0] | 6.3 [4.5 to 8.2]
Statistical Analysis 1: Comparison: Sunitinib (Phase 3) vs Imatinib; Test type: Superiority or Other; Cox Proportional Hazards Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.027, 95% CI 2-sided [0.505 to 2.088]

5. Secondary Outcome: Number of Participants With Objective Response of Complete Response or Partial Response
Description: Number of participants with objective response based assessment of confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as the disappearance of all target lesions. PR was defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 31 | 26
Participants | 5 | 2
Statistical Analysis 1: Comparison: Sunitinib (Phase 3) vs Imatinib; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Stratified by previous imatinib treatment status (less than 6 months of treatment with imatinib and greater than or equal to 6 months); Odds Ratio (OR) = 2.308, 95% CI 2-sided [0.4 to 13.0]

6. Secondary Outcome: Time to Tumor Response (TTR)
Description: Time from date of randomization to first documentation of objective tumor response (partial or complete response). Confirmed complete response (CR) and partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as the disappearance of all target lesions. PR was defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 31 | 26
Weeks | 4.1 [3.6 to 20.1] | 40.1 [5.4 to 74.7]

7. Secondary Outcome: Duration of Response (DR)
Description: Time from start of first documentation of objective response(complete or partial response) that was subsequently confirmed to first documentation of objective tumor progression or death due to any cause, whichever occurred first.
  Confirmed complete response (CR) and partial response (PR)according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as the disappearance of all target lesions. PR was defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT; Number of participants analyzed: participants with an objective tumor response. DR data censored on the day following the date of the last tumor assessment on study for participants who did not have objective tumor progression and who did not die due to any cause while on study.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 5 | 2
Weeks | 18.3 [7.9 to 24.1] | 19.8 [6.7 to 32.9]

8. Secondary Outcome: Time to Pain Progression (TTPP)
Description: TTPP is the number of days from randomization to the first documentation of pain progression (defined as a 50% or more increase in MPQ-PPI score [0=no pain to 5=excruciating pain] or analgesic use from baseline for at least 3 consecutive weeks). Analgesic use scores were based on 1 point per non narcotic dose of medication and 4 points per dose of narcotic medication.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT; Number of participants analyzed: participants with an event.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 14 | 10
Days | 22.0 [8.0 to 29.0] | 99.0 [8.0 to 134.0]
Statistical Analysis 1: Comparison: Sunitinib (Phase 3) vs Imatinib; Test type: Superiority or Other; Cox Proportional Hazards Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 3.434, 95% CI 2-sided [1.057 to 11.15]

9. Secondary Outcome: Number of Participants With Pain Relief Response
Description: Pain relief response defined as a 50% or more reduction in the McGill Pain Questionaire - Present Pain Intensity (MPQ-PPI) score (0=no pain to 5=excruciating pain) and/or analgesic use from baseline for at least 3 consecutive weeks. Analgesic use scores were based on 1 point per non narcotic dose of medication and 4 points per dose of narcotic medication.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT; Number of participants analyzed: participants with MPQ-PPI and analgesic use data at baseline.
Measure: Number; unit: Participants
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 7 | 10
Participants | 2 | 4
Statistical Analysis 1: Comparison: Sunitinib (Phase 3) vs Imatinib; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Stratified for previous imatinib treatment status (less than 6 months of treatment with imatinib and greater than or equal to 6 months); Odds Ratio (OR) = 0.379, 95% CI 2-sided [0.1 to 2.3]

10. Secondary Outcome: Number of Participants With Pain Progression
Description: Pain progression defined as a 50% or more increase in MPQ-PPI score (0=no pain to 5=excruciating pain) or analgesic use from baseline for at least 3 consecutive weeks. Analgesic use scores were based on 1 point per non narcotic dose of medication and 4 points per dose of narcotic medication.
Time Frame: Day 28 of Cycle 1 up to 26
Population: ITT; Number of participants analyzed: participants with MPQ-PPI and analgesic use data at baseline.
Measure: Number; unit: Participants
Arm/Group | Sunitinib (Phase 3) | Imatinib
Number analyzed (Participants) | 23 | 21
Participants | 14 | 10
Statistical Analysis 1: Comparison: Sunitinib (Phase 3) vs Imatinib; Test type: Superiority or Other; Cochran-Mantel-Haenszel; [statistical method as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.318, 95% CI 2-sided [0.5 to 3.8]

11. Secondary Outcome: Euro Quality of Life (EQ-5D) - Health State Profile Utility Score- Sunitinib Treatment Arm
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component rated current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicated better health state (no problems); 3 indicated worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigned utility value for each domain in profile. Score was transformed and results in a total score ranged 0.21 to 1.000; higher score indicated a better health state.
Time Frame: Days 1 and 28 of each cycle
Population: ITT; Number of participants analyzed: participants who completed the scale; n: participants who completed the scale at the respective cycle.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sunitinib (Phase 3)
Number analyzed (Participants) | 30
Scores on a scale
  Cycle 1 (n=30) | 0.90 (0.159)
  Cycle 2 (n=27) | 0.84 (0.196)
  Cycle 3 (n=21) | 0.84 (0.130)
  Cycle 4 (n=23) | 0.85 (0.186)
  Cycle 5 (n=16) | 0.89 (0.133)
  Cycle 6 (n=16) | 0.90 (0.120)
  Cycle 7 (n=12) | 0.84 (0.182)
  Cycle 8 (n=11) | 0.83 (0.168)
  Cycle 9 (n=6) | 0.76 (0.149)
  Cycle 10 (n=5) | 0.78 (0.128)
  Cycle 11 (n=3) | 0.83 (0.157)
  Cycle 12 (n=2) | 0.93 (0.106)

12. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS) - Sunitinib Treatment Arm
Description: EQ-5D: participant rated questionnaire assessed health-related quality of life in terms of a single index value. The VAS component rated current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicated a better health state.
Time Frame: Days 1 and 28 of each cycle
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Sunitinib (Phase 3)
Number analyzed (Participants) | 30
Scores on a Scale
  Cycle 1 (n=30) | 78.13 (23.80)
  Cycle 2 (n=27) | 77.19 (19.98)
  Cycle 3 (n=21) | 78.52 (14.24)
  Cycle 4 (n=23) | 80.17 (14.28)
  Cycle 5 (n=16) | 84.25 (12.30)
  Cycle 6 (n=16) | 85.81 (13.25)
  Cycle 7 (n=12) | 78.25 (15.91)
  Cycle 8 (n=11) | 84.73 (12.71)
  Cycle 9 (n=7) | 82.57 (14.30)
  Cycle 10 (n=6) | 81.00 (12.59)
  Cycle 11 (n=3) | 81.00 (14.93)
  Cycle 12 (n=2) | 86.50 (16.26)

13. Secondary Outcome: Euro Quality of Life (EQ-5D) - Health State Profile Utility Score - Imatinib Treatment Arm
Description: EQ-5D: participant rated questionnaire assessed health-related quality of life in terms of a single utility score. Health State Profile component rated current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicated better health state (no problems); 3 indicated worst health state (eg, "confined to bed"). Scoring formula developed by EuroQol Group assigned utility value for each domain in the profile. Score was transformed and results in a total score ranged 0.21 to 1.000; higher score indicated a better health state.
Time Frame: Days 1 and 28 of each cycle
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Imatinib
Number analyzed (Participants) | 23
Scores on a scale
  Cycle 1 (n=22) | 0.80 (0.117)
  Cycle 2 (n=23) | 0.85 (0.135)
  Cycle 3 (n=18) | 0.82 (0.162)
  Cycle 4 (n=18) | 0.86 (0.143)
  Cycle 5 (n=17) | 0.83 (0.217)
  Cycle 6 (n=12) | 0.84 (0.157)
  Cycle 7 (n=12) | 0.81 (0.260)
  Cycle 8 ( (n=11) | 0.68 (0.292)
  Cycle 9 (n=7) | 0.86 (0.105)
  Cycle 10 (n=7) | 0.86 (0.104)
  Cycle 11 (n=3) | 0.88 (0.106)

14. Secondary Outcome: Euro Quality of Life (EQ-5D)- Visual Analog Scale (VAS) - Imatinib Treatment Arm
Description: as for outcome 12
Time Frame: Days 1 and 28 of each cycle
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Imatinib
Number analyzed (Participants) | 22
Scores on a scale
  Cycle 1 (n=22) | 75.41 (16.60)
  Cycle 2 (n=22) | 73.64 (14.61)
  Cycle 3 (n=20) | 72.85 (15.24)
  Cycle 4 (n=18) | 76.14 (15.78)
  Cycle 5 (n=15) | 68.93 (12.82)
  Cycle 6 (n=11) | 68.27 (15.10)
  Cycle 7 (n=12) | 67.08 (18.08)
  Cycle 8 (n=10) | 63.70 (19.23)
  Cycle 9 (n=7) | 74.64 (13.26)
  Cycle 10 (n=7) | 76.86 (8.009)
  Cycle 11 (n=3) | 75.33 (5.508)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. One participant enrolled in the imatinib arm was inadvertently randomized (participant did not meet inclusion criteria) and was not treated in this study.
Groups:
- All Participants Who Received Sunitinib: Participants in Phase 1 sub- study and Phase 3 study
- Imatinib: All participants who received Imatinib
Arm/Group | All Participants Who Received Sunitinib | Imatinib
Serious Adverse Events (participants affected / at risk) | 11/43 | 5/25
Other Adverse Events (participants affected / at risk) | 43/43 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants Who Received Sunitinib (N=43) | Imatinib (N=25)
Myocardial infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Disease progression (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants Who Received Sunitinib (N=43) | Imatinib (N=25)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 0
Hypothyroidism (Endocrine disorders) | 3 | 1
Eyelid oedema (Eye disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhoea (Gastrointestinal disorders) | 19 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 1
Flatulence (Gastrointestinal disorders) | 3 | 0
Glossodynia (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 12 | 9
Oral pain (Gastrointestinal disorders) | 3 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 6 | 6
Asthenia (General disorders) | 5 | 2
Face oedema (General disorders) | 1 | 2
Fatigue (General disorders) | 13 | 8
Feeling cold (General disorders) | 0 | 2
Mucosal inflammation (General disorders) | 15 | 0
Oedema (General disorders) | 0 | 5
Oedema peripheral (General disorders) | 4 | 5
Pyrexia (General disorders) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Dysgeusia (Nervous system disorders) | 9 | 0
Headache (Nervous system disorders) | 6 | 2
Lethargy (Nervous system disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1
Blister (Skin and subcutaneous tissue disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Hair colour changes (Skin and subcutaneous tissue disorders) | 3 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 4
Yellow skin (Skin and subcutaneous tissue disorders) | 3 | 0
Flushing (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 16 | 0

LIMITATIONS AND CAVEATS:
On 18 June 2009, the study was prematurely stopped for operational reasons (poor recruitment, lack of interest, and change of clinical practice) and not related to safety concerns

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.